CLINICAL TRIAL: NCT07306013
Title: The SolanoConnex Trial: A Single-blind Randomized Controlled Trial of a Digital and Community-based Mental Health Access Project
Brief Title: The SolanoConnex Trial: Evaluation of a Mental Health Access Project
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Touro University, California (Other)
Collaborators: Solano County Board of Supervisors (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MHAS2025
Record Dates: First submitted 2025-07-14; First posted 2025-12-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Mental Health
Keywords: mental health; web application; community-based
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mental Health Navigator and App Intervention Group (Experimental): Participants in the intervention group will be blinded to their study arm status. They will receive full access and orientation to SolanoConnex.org, including multiple features designed to enhance engagement with local mental health resources. First, they will be granted access to the SolanoConnex.org website and mobile application, educational materials, social media and resource navigation. To facilitate ease of use, participants will receive a step-by-step guide and a tutorial video demonstrating how to navigate the platform's features. Additionally, they will gain access to SolanoConnex-produced videos and podcasts which profiles mental health providers and covers various mental health topics.
  Interventions: Behavioral: Access to the SolanoConnex.org
- Standard County Mental Health Information Control (No Intervention): Participants in the control group will also be blinded to their study arm status. They will receive generic materials consisting of access to publicly available mental health resources without exposure to SolanoConnex.org or its patient navigator services. They will be provided with general information on national mental health hotlines, local mental health services, and online directories of available resources but will not receive specific training or guidance in using these resources.

INTERVENTIONS:
Behavioral: Access to the SolanoConnex.org — Participants in the intervention group will be blinded to their study arm status. They will receive full access and orientation to SolanoConnex.org, including multiple features designed to enhance engagement with local mental health resources.
  First, they will be granted access to the SolanoConnex.org website and mobile application, educational materials, social media and resource navigation. To facilitate ease of use, participants will receive a step-by-step guide and a tutorial video demonstrating how to navigate the platform's features. Additionally, they will gain access to SolanoConnex-produced videos and podcasts which profiles mental health providers and covers various mental health topics.
  To further support participants, patient navigators will be available to provide personalized assistance, helping individuals connect with relevant services. At the outset of the study, participants will receive detailed instructions on how to access and utilize patient navigator support.
  Arms: Mental Health Navigator and App Intervention Group

SUMMARY:
The goal of this study is to evaluate the effectiveness of the SolanoConnex.org program on help-seeking attitudes and help-seeking behaviors among users compared to a control group. This study will employ a randomized controlled trial design with two parallel arms. Participants in the intervention group will receive full access and orientation to SolanoConnex.org, including multiple features designed to enhance engagement with local mental health resources. Participants in the control group will receive publicly available mental health resources. The primary outcome is any use of mental health services including conversations and communication, digital engagement and media consumption, direct service use or self-help and alternative support all of which will be self-reported through digital diaries prompted every two weeks. Secondary outcomes are endorsed and anticipated Stigma related to mental health, help-seeking attitudes, self-efficacy in seeking mental health care. Potential covariates include demographics, past mental health service use and satisfaction, readiness to change, and discrimination experiences during past healthcare use.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Resident of Solano County, CA.
* Mild to moderate mental health symptoms as reported on the DSM-5 Level 1 Measure for Adult Mental Health screening form.
* Own a personal smartphone with internet access or a data plan to facilitate engagement with the digital platform.
* Be fluent in English, as all study components will be conducted in English.
* Have not previously used SolanoConnex.org.

Exclusion Criteria:

* Are currently engaged in or have had comprehensive case management or counseling services within the past 6 months.
* Do not reside in Solano County.
* Lack fluency in English, as study materials and communications will be conducted in English.
* Have previously accessed SolanoConnex.org, as prior exposure may influence study outcomes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-07-13 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Use of any mental health services | From enrollment to the end of the 4 month study period
  Mental health service utilization (i.e. appointment with therapist, attendance at grief group, commencement of PTSD treatment)

SECONDARY OUTCOMES:
Stigma Related to Mental Health | From enrollment to the end of the 4 month period
  Endorsed and Anticipated Stigma Inventory (EASI): The EASI is a 40-item self-report inventory that consists of 5 scales assessing mental health beliefs that may be particularly salient for military and Veteran populations, particularly with regard to their willingness to seek mental health treatment. Respondents are asked to rate 8 items in each of 5 scales, 3 that address key aspects of endorsed stigma and 2 that assess key aspects of anticipated stigma. Each scale uses a 5-point Likert-type response format: 1 (strongly disagree), 2 (somewhat disagree), 3 (neither agree nor disagree), 4 (somewhat agree), 5 (strongly agree). Items within each of the 5 scales can be summed to create individual 5 scale scores. The higher the score, the higher the stigma.
Mental Health Help Seeking Attitudes | From enrollment to the end of the 4 month period
  Mental Help Seeking Attitudes Scale (MHSAS): The MHSAS contains nine items which produce a single mean score. The MHSAS uses a seven-point semantic differential scale. In order to properly calculate the MHSAS mean score, where a higher mean score indicates more favorable attitudes, it is necessary to reverse-code items 2, 5, 6, 8, and 9.
Self-efficacy in seeking Mental Health Care | From enrollment to the end of the 4 month period
  Self-efficacy in Seeking Mental Health Care Scale: Sum all 9 items. Higher scores indicate greater self-efficacy for seeking mental health care.

CONTACTS AND LOCATIONS:
Locations (1):
- Touro University, California, Vallejo, California, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD), including the analyzable dataset underlying published results, may be shared.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: July 1 2026 - June 31, 2027
Access Criteria: De-identified IPD will be made available upon reasonable request to qualified researchers, subject to approval by the study investigators and completion of a data use agreement. Requests should specify the research question, analysis plan, and intended use of the data.

REFERENCES:
- See also: Recruitment site — http://www.SolanoMentalHealthStudy.org